CLINICAL TRIAL: NCT06581198
Title: A Phase 2, Open-label, Study to Evaluate the Efficacy and Safety of Rapcabtagene Autoleucel in Patients With Active, Refractory Systemic Lupus Erythematosus (SLE) or Active, Refractory Lupus Nephritis (LN).
Brief Title: A Study of Rapcabtagene Autoleucel in Active, Refractory Systemic Lupus Erythematosus (SLE) or Lupus Nephritis (LN) Patients (AUTOGRAPH - SLE/LN)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CYTB323J12201; 2023-510150-17-00 (Registry Identifier: EU CT Number)
Record Dates: First submitted 2024-08-23; First posted 2024-09-03 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Lupus Erythematosus, Systemic; Lupus Nephritis
Keywords: Chimeric Antigen Receptor-T (CAR-T); rapcabtagene autoleucel; Lupus Nephritis (LN); Systemic Lupus Erythematosus (SLE)
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Lupus Nephritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- rapcabtagene autoleucel (Experimental): rapcabtagene autoleucel
  Interventions: Biological: rapcabtagene autoleucel

INTERVENTIONS:
Biological: rapcabtagene autoleucel — single infusion of rapcabtagene autoleucel

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of rapcabtagene autoleucel (administered once following lymphodepletion) in patients with active, refractory systemic lupus erythematosus (SLE) or active, refractory lupus nephritis (LN).

ELIGIBILITY:
Key Inclusion Criteria:

* Men and women with SLE, aged >= 18 years and =< 75 years at screening, fulfilling the 2019 European League Against Rheumatism (EULAR)/American College of Rheumatology (ACR) classification criteria for SLE at screening.
* Participant must be positive for at least one of the following autoantibodies at screening: antinuclear antibodies (ANA) at a titer of >= 1:80 (on HEp-2 cells or an equivalent positive test), or anti-dsDNA (above the ULN); or anti-Sm (above the ULN) as determined by a central laboratory.
* Active lupus nephritis without signs of significant chronicity or active systemic lupus erythematosus
* SLEDAI-2K Criteria at screening: SLEDAI-2K score >= 6 points (Gladman et al 2002, Touma et al 2011), excluding points attributed to "fever", "lupus headache", "alopecia", and "organic brain syndrome".
* Inadequate response at screening to at least two therapies

Key Exclusion Criteria:

* Any acute, severe lupus related-flare at screening that needs immediate treatment other than pulse GCs and/or makes the immunosuppressive washout impossible and, thus, makes the participant ineligible for CD19 CAR-T therapy
* Inadequate organ function during screening and prior to randomization
* History or current diagnosis of ECG or cardiac abnormalities indicating significant risk of safety for participants prior to randomization
* Human immunodeficiency virus (HIV) positivity at screening.
* Acute or chronic infection with hepatitis B (HBV) or hepatitis C (HCV) at screening.
* Grade 2 or higher thromboembolic event in the past 4 weeks prior to screening.

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 179 (Estimated)
Dates: Start 2024-09-04 (Actual); Primary Completion 2028-02-14 (Estimated); Study Completion 2032-02-06 (Estimated)

PRIMARY OUTCOMES:
Evaluate the efficacy of rapcabtagene autoleucel | Week 24, Week 52
  Defined as:
  Meeting the criteria of the Definition Of Remission In Systemic Lupus Erythematosus (DORIS)
  or
  Achieving complete renal response (CRR)

SECONDARY OUTCOMES:
Percentage of participants achieving complete renal response (CRR) | Week 52
  CRR is a composite endpoint
Number of weeks where Lupus Low Disease Activity Score (LLDAS) was achieved | Week 12 to Week 52
  Lupus Low Disease Activity State (LLDAS)
PPercentage of participants without flaring (i.e., 1 new BILAG2004 A or 2 new BILAG2004 B flares) | Week 12 to Week 52
  British Isles Lupus Activity Group (BILAG2004) records disease activity occurring over the past 4 weeks.
Annualized cumulative corticosteroids dose | Week 52
  The total dose of corticosteroids used up to Week 52 per patient.
Percentage of participants who are negative for serological status | Week 52
  The percentage of participants with negative serological status
FACIT-Fatigue score change from baseline | Baseline to Week 52
  Functional Assessment of Chronic Illness Therapy (FACIT)-Fatigue is a 13-item patient- reported outcomes measure
Maintained DORIS | Week 52 to Week 76
  Definition Of Remission In Systemic Lupus Erythematosus (DORIS)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (81):
- United States (15):
  - University Of Alabama, Birmingham, Alabama
  - Loma Linda University, San Bernardino, California
  - UCSF, San Francisco, California
  - Sutter Health Network, San Pablo, California
  - Ann and Robert H Lurie Childs Hosp, Chicago, Illinois
  - Northwestern University, Chicago, Illinois
  - University Of Iowa, Iowa City, Iowa
  - University of Kentucky, Lexington, Kentucky
  - Tufts Medical Center, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - WA Uni School Of Med, St Louis, Missouri
  - Oregon Health Sciences University, Portland, Oregon
  - Univ Of TX MD Anderson CC, Houston, Texas
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - LDS Hospital, Salt Lake City, Utah
- Novartis Investigative Site, Clayton, Victoria, Australia
- Austria (2):
  - Novartis Investigative Site, Graz
  - Novartis Investigative Site, Vienna
- Brazil (3):
  - Novartis Investigative Site, Salvador, Estado de Bahia
  - Novartis Investigative Site, São Paulo, São Paulo
  - Novartis Investigative Site, São Paulo
- Czechia (2):
  - Novartis Investigative Site, Olomouc
  - Novartis Investigative Site, Prague
- Novartis Investigative Site, Aarhus N, Denmark
- France (6):
  - Novartis Investigative Site, Bordeaux
  - Novartis Investigative Site, Marseille
  - Novartis Investigative Site, Nantes
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Toulouse
  - Novartis Investigative Site, Vandœuvre-lès-Nancy
- Germany (9):
  - Novartis Investigative Site, Stuttgart, Baden-Wurttemberg
  - Novartis Investigative Site, Frankfurt am Main, Hesse
  - Novartis Investigative Site, Cologne, North Rhine-Westphalia
  - Novartis Investigative Site, Leipzig, Saxony
  - Novartis Investigative Site, Jena, Thuringia
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Mainz
  - Novartis Investigative Site, Nuremberg
  - Novartis Investigative Site, Ulm
- Hungary (2):
  - Novartis Investigative Site, Debrecen, Hajdu Bihar Megye
  - Novartis Investigative Site, Budapest
- Italy (6):
  - Novartis Investigative Site, Ancona, AN
  - Novartis Investigative Site, Genova, GE
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Rozzano, MI
  - Novartis Investigative Site, Pisa, PI
  - Novartis Investigative Site, Pavia, PV
- Japan (12):
  - Novartis Investigative Site, Sapporo, Hokkaido
  - Novartis Investigative Site, Kobe, Hyōgo
  - Novartis Investigative Site, Kanazawa, Ishikawa-ken
  - Novartis Investigative Site, Yokohama, Kanagawa-ku
  - Novartis Investigative Site, Sendai, Miyagi
  - Novartis Investigative Site, Suita, Osaka
  - Novartis Investigative Site, Izumo, Shimane
  - Novartis Investigative Site, Bunkyo Ku, Tokyo
  - Novartis Investigative Site, Bunkyo-ku, Tokyo
  - Novartis Investigative Site, Chiba
  - Novartis Investigative Site, Fukuoka
  - Novartis Investigative Site, Kyoto
- Netherlands (3):
  - Novartis Investigative Site, Leiden, South Holland
  - Novartis Investigative Site, Groningen
  - Novartis Investigative Site, Utrecht
- Novartis Investigative Site, Oslo, Norway
- Novartis Investigative Site, Bucharest, Romania
- Novartis Investigative Site, Riyadh, Saudi Arabia
- Novartis Investigative Site, Singapore, Singapore
- Novartis Investigative Site, Seoul, South Korea
- Spain (8):
  - Novartis Investigative Site, Santiago Compostela, A Coruna
  - Novartis Investigative Site, Santander, Cantabria
  - Novartis Investigative Site, Pamplona, Navarre
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Córdoba
  - Novartis Investigative Site, Madrid
  - Novartis Investigative Site, Salamanca
  - Novartis Investigative Site, Valencia
- Novartis Investigative Site, Stockholm, Sweden
- Novartis Investigative Site, Lausanne, Switzerland
- Taiwan (2):
  - Novartis Investigative Site, Taichung
  - Novartis Investigative Site, Taipei
- United Kingdom (2):
  - Novartis Investigative Site, Sheffield, South Yorkshire
  - Novartis Investigative Site, London

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations. This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com.
URL: https://www.clinicalstudydatarequest.com